CLINICAL TRIAL: NCT06677905
Title: SCI&U Peer Health Coaching Program for Individuals Newly Discharged From Inpatient Rehabilitation
Acronym: SCIU2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Susan Jaglal, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 977608
Record Dates: First submitted 2024-11-04; First posted 2024-11-07 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury
Keywords: peer support; self-management; spinal cord injury; newly injured; web-based program
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCI&U self-management program (Experimental): Following recruitment intervention participants will be scheduled for an orientation session to become better acquainted with the health coaching program and the associated platform's features. Participants will then be partnered with their peer health coach. In the first videoconference session, participants will identify priority issues related to their health and transitioning to home. They will work through goal-setting, problem solving and create action plans for behaviour change. Online coaching sessions are expected to cover a health-related topic and a self-management skill topic and will have an expected duration of 45 to 60 minutes. The selection of topics and the order will be determined jointly.
  Interventions: Behavioral: web-based spinal cord injury self-management program
- Wait list control (Active Comparator): Control group will be offered the existing peer support program from the United Spinal Connecticut Chapter or SCI BC
  Interventions: Behavioral: Peer support

INTERVENTIONS:
Behavioral: web-based spinal cord injury self-management program — Peer health coaches will be recruited from the United Spinal Connecticut Chapter and SCI BC. They will be at least 5 years post-SCI and will be certified in brief action planning and in Mental Health First Aid.
  Online coaching sessions are expected to cover a health-related topic (eg. bladder, bowel, skin, pain, healthy eating, physical activity or stress, anxiety and depression etc) and a self-management skill topic (eg.action planning, goal setting, problem-solving, mood management, navigating the health care system, communicating with health care providers). To ensure we meet the unique needs of participants, the coach and participant will determine jointly how many sessions to spend on a topic. In addition, coaches will be able to link relevant information and resources contained in the resource library to each session.
  Arms: SCI&U self-management program
Behavioral: Peer support — Existing peer support program from the United Spinal Connecticut Chapter or SCI BC
  Arms: Wait list control

SUMMARY:
The goal of this clinical trial is to learn if the online program and web-based platform for delivery of self-management services to people with spinal cord injury (SCI) called "SCI & U" can support transitions from hospital to the community after injury. Specifically, can providing support from trained peer health coaches via the SCI & U web-based self-management program increase health self-management among those within three years of a spinal cord injury with a planned discharge to or living in the community with SCI for less than two years in the province of British Columbia, Canada or the state of Connecticut, United States.

The main question it aims to answer is:

• Does the SCI & U web-based self-management program lower emotional distress and increase self-efficacy Researchers will compare those who participate in SCI & U with those who receive usual peer support after 6 months to see if the SCI & U program improves self-management knowledge, skills and self-efficacy and decreases secondary complications

Participants will:

* engage in up to 14 online sessions, each of which lasts about an hour with a peer health coach trained in motivational interviewing, goal setting and brief action planning. During sessions, they may also review resources and create follow up plans on the online platform on health management topics
* complete an interviewer administered survey at baseline, 6 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older, with a planned discharge to or living in community with SCI for no more than three years since injury and with the ability to speak and understand English

Exclusion Criteria:

* not a member of or willing to become a member of SCI BC or SCIACT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Emotional Distress Subscale in Health Education Impact Questionnaire | From baseline assessment to 6 months followup
  The Emotional Distress construct measures overall negative affect including worry, depression and anger.

SECONDARY OUTCOMES:
Health Directed Activities in Health Education Impact Questionnaire | From baseline assessment to 6 months followup
Positive and Active Engagement in Life in Health Education Impact Questionnaire | From baseline assessment to 6 months followup
Self-monitoring and Insight in Health Education Impact Questionnaire | From baseline assessment to 6 months followup
Constructive Attitudes and Approaches in Health Education Impact Questionnaire | From baseline assessment to 6 months followup
Skill and Technique Acquisition in Health Education Impact Questionnaire | From baseline assessment to 6 months followup
Social Integration and Support in Health Education Impact Questionnaire | From baseline assessment to 6 months followup
Health Services Navigation in Health Education Impact Questionnaire | From baseline assessment to 6 months followup
The Patient Activation Measure - (PAM) Survey | From baseline assessment to 6 months followup
  The Patient Activation Measure (PAM) is a commercial product which assesses an individual's knowledge, skill, and confidence for managing one's health and healthcare. The PAM survey measures patients on a 0-100 scale and can segment patients into one of four activation levels. Individuals who measure high on this assessment typically understand the importance of taking a pro-active role in managing their health and have the skills and confidence to do so.
Moorong Self-Efficacy Scale | From baseline assessment to 6 months followup
  Measures self-efficacy in performing functional activities of daily living in individuals with SCI.
  Consists of two factors: daily activities (e.g., I can maintain my personal hygiene with or without help), and social functioning (e.g., I can enjoy spending time with my friends)
Secondary Conditions Scale | From baseline assessment to 6 months followup
  A 16-item self-report measure that targets secondary conditions associated with SCI that impact health on a 4-point scale from "not experienced in the last 3 months" to significant or chronic problem"
NIH Toolbox Loneliness Scale | From baseline assessment to 6 months followup
System Usability Scale | From baseline assessment to 6 months followup
  This scale was designed to evaluate the usability of interactive systems flexibly and expediently.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Jaglal, PhD, Principal Investigator — University of Toronto
Locations (2):
- Spinal Cord Injury Association of Connecticut, Milford, Connecticut, United States
- Department of Physical Therapy, University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared only for those who consent to their data being shared. The data will be deposited into a database. Any information that may identify an individual (e.g., name, address, phone number) will not be shared. In addition to data on outcome measures, descriptive variables and covariates, data describing participation in the intervention also will be shared. This will include number of sessions participants completed, length of sessions, topics discussed and if brief action plan was developed and goals set.
Supporting Information: SAP, ICF
Time Frame: IPD will be available in January 2028 which provides 1 year for publication of the main study results in a peer-reviewed journal article
Access Criteria: We will make the content available publicly. This will include analytic datasets with data on outcome measures, descriptive variables and covariates and data describing participation in the intervention. Supporting information including the SAP and ICF will also be made available. Data will be deposited in the University of Toronto Dataverse which is a research data repository. Files will held in a secure environment on Canadian servers.